CLINICAL TRIAL: NCT04847076
Title: Preliminary Evaluation of the Effectiveness of the Intervention And Now What? to Promote Maternal Mental Health in the Postpartum Period in the Primary Health System in Chile.
Brief Title: Feasibility of M-health Version of "What Were We Thinking" Intervention to Promote Maternal Postpartum Mental Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad del Desarrollo (Other)
Collaborators: Instituto Milenio para Investigación en Depresión y Personalidad (Other); Peñalolén County Corporation, Chile (Unknown)
Responsible Party: Principal Investigator, Soledad Coo Calcagni, Faculty of Psychology, Universidad del Desarrollo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MIDAP2020FIP1
Record Dates: First submitted 2021-04-05; First posted 2021-04-15 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Depression, Postpartum; Anxiety Disorders and Symptoms; Maternal Behavior
Keywords: Feasibility Studies; Prevention; mHealth
MeSH Terms: conditions — Depression, Postpartum; Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to intervention or control groups at a 1:1 ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- m-health version of WWWT intervention (Experimental): Include: a) Psychoeducational information for understanding and managing infant behavior and on parenting. This information will be delivered through instant messaging service for mobile phones (i.e., Whatsapp) 3 times a week for four-week period. Each module will include a very brief video offering information regarding a specific topic, a proposed personal exercise and the invitation to assess the perceived usefulness of the information received. Some modules include links to external, complementary information from the Chilean Infancy Policy. b) Contact with the program facilitator. It will allow mothers to ask questions that arise from the topics addressed in the psychoeducational videos. The answers seek to promote the understanding and elaboration of the contents, and operate by providing expert support; c) A virtual group meeting.
  Interventions: Behavioral: m-health version of WWWT intervention
- TREATMENT AS USUAL (Other): TAU for children under one year of age include routine health checks by health professionals (nurse or doctor), every month from 0 to 4 months of age, and at 6, 8 and 12 months of age. The objective of the routine health care check is to carry out a comprehensive evaluation of the child's development and growth, guide parents and caregivers regarding child development, health and upbringing of the child. Also, promoting exclusive breastfeeding, healthy mother/child bonding (by detecting relevant alterations in this area) and encouraging paternal participation in upbringing and care of the child. Finally, in the health check-ups at 2 and 6 months of age of the child, Edinburgh Postpartum Depression Scale is used for screening depressive symptoms in mothers. At risk cases are referred for mental health assessment and care.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: m-health version of WWWT intervention — m-health version of Chilean adaptation of WWWT intervention: a) Psychoeducational information for understanding and managing infant behavior and on parenting. b) Contact with the program facilitator. c) A virtual group meeting
  Arms: m-health version of WWWT intervention
Other: Treatment as usual — TAU for children under one year of age include routine health checks by health professionals (nurse or doctor), every month from 0 to 4 months of age, and at 6, 8 and 12 months of age
  Arms: TREATMENT AS USUAL

SUMMARY:
The purpose of this study is to assess the feasibility, acceptability and preliminary effectiveness of "What Were We Thinking" (WWWT) a psychoeducational intervention -delivered remotely via communication technologies- to prevent symptoms of postpartum depression and anxiety in new mothers; which has been shown to be effective in primary health settings. WWWT was developed in Australia and has been culturally adapted to be used in Chile. The m-health version of the Chilean adaptation of WWWT for the current study includes: Psychoeducational modules on issues relevant to mothers during the post-partum period; contact with the program facilitator through instant messaging services available on mobile phones and a virtual group meeting.

This pilot study will use a mixed design. The quantitative component will consist of a before-after design with control group including 90 adult mothers of child aged 6-8 weeks who receive health care in a primary health centers in Santiago, Chile. Mothers will be randomized into the experimental (EG) or control groups (CG) in a rate of 1:1. Both EG and CG will receive usual treatment provided by primary health centers (TAU), and only de EG will receive the m-health adapted version of the WWWT.

The qualitative component considers 12 users semi-structured interviews. The maximum variation sampling strategy will be used according to the completion of m-health version of WWWT. An open coding of Grounded Theory will be used to data analysis.

The feasibility of m-health version of WWWT intervention will be evaluated in terms of eligibility rates, recruitment rates and reasons for study refusals, feasibility to deliver the three components of the intervention, data attrition and follow-up rates by treatment condition. Their acceptability considers participant completion of the intervention rates, and a qualitative assessment of the users' acceptability of and satisfaction. Secondary outcomes will include changes on maternal levels of depressive and anxiety symptoms, maternal self-efficacy and perceived social support. And differences in mother-infant quality of interaction between intervention and control groups.

DETAILED DESCRIPTION:
Mental health symptoms are common in new mothers. Despite the availability of effective screening and referral in the primary health system in Chile, very few women access treatment due to diverse barriers (i.e., long waiting lists and insufficient knowledge about postnatal depression and treatment). This highlights the importance of using a preventive approach. Currently in Chile there are no universal preventive interventions, although they are available internationally.

Thus, this study seeks to assess if it's feasible and acceptable to offer an alternative intervention that can be delivered remotely by mobile phones, to support women in the early postpartum period by promoting confidence and reducing distress in first time mothers. By doing so, it will increase the number of available interventions to promote and prevent children´s early adverse experiences related to maternal mental health problems.

This study accounts for the feasibility, acceptability and preliminary effectiveness of "What Were We Thinking" (WWWT) a psychoeducational intervention -delivered remotely via communication technologies- to prevent symptoms of postpartum depression and anxiety in new mothers. WWWT was developed in Australia and has been culturally adapted to be used in Chile. The m-health version of the Chilean adaptation of WWWT includes:

1. Psychoeducational information for understanding and managing infant behavior and about parenting. Modules on understanding and managing infant behavior include information on: infant temperament, including such as differences in the reactivity, responsivity and regulation of young infants; amount and known and unknown reasons for infant crying; stimulation, over-stimulation and soothing; infant sleep needs and optimal sleep habits; the use of settling strategies to achieve these while supporting breastfeeding; and establishing sustainable routines of daily care: the feed, play, sleep routine. Modules on matters relating to parents include: gendered differences in the losses and gains of parenthood; differences in emotional needs and the potential for adverse reproductive events to have lasting psychological effects on women after the birth of a baby; and developing strategies to assist couples to address these in a non-confrontational manner. This information will be delivered through instant messaging services for mobile phones (i.e., Whatsapp) 3 times a week for four-week period. Each module will include a very brief video offering information regarding a specific topic, a proposed personal exercise and the invitation to assess the perceived usefulness of the information received. Some modules include links to external, complementary information from the Chilean Infancy Policy.
2. Contact with the program trained facilitator. It will allow mothers to ask questions that arise from the topics addressed in the psychoeducational videos and share their personal experiences. The facilitator responses will focus on aiding the understanding and elaboration of the contents. This will be done through instant messaging service for mobile phones (i.e., Whatsapp). In the present study, the facilitator will be a mental health professional of the research team, that has been trained on the intervention model.
3. Group virtual meeting. A virtual group meeting will take place with mothers and their partners (or significant others) and the program facilitator. The group meeting seeks to offer an instance were new mothers and fathers can share their experiences regarding their parenthood and the changes it has involved in their daily lives, as well as providing the opportunity for developing support networks among them.

This pilot study will use a mixed design. The quantitative component will consist of a before-after design with control group including 90 adult mothers of child aged 6-8 weeks who receive health care in a primary health centers in Santiago. Mothers will be randomized into the experimental (EG) or control groups (CG) in a rate of 1:1. Mothers in the EG will receive the m-health version of WWWT intervention plus the usual treatment that primary health centers (TAU) provided to children. Participants in the CG will be subject to TAU. TAU for children under one year of age include routine health checks by health professionals (nurse or doctor), every month from 0 to 4 months of age, and at 6, 8 and 12 months of age. The objective of the routine health care check is to carry out a comprehensive evaluation of the child's development and growth, guide parents and caregivers regarding child development, health and upbringing of the child. Also, promoting exclusive breastfeeding, healthy mother/child bonding (by detecting relevant alterations in this area) and encouraging paternal participation in upbringing and care of the child. Finally, in the health check-ups at 2 and 6 months of age of the child, Edinburgh Postpartum Depression Scale is used for screening depressive symptoms in mothers. At risk cases are referred for mental health assessment and care. A waiting list procedure will allow the delivery of the intervention to control women once the data collection for the study has been completed.

The participating mothers will be contacted in coordination with the health providers of two public primary health centers after the first newborn health check. All women who meet the inclusion criteria will be contacted by the research assistant to participate of the research project. Women who wish to participate will be randomly assigned to the EG or CG. Both groups will receive informed consent and will be assessed regarding sociodemographic characteristics, mother's symptoms of anxiety and depression, maternal self-efficacy and perceived social support. The participants in both groups will be assessed a week before the start of the intervention (baseline) and three months after its completion (follow-up). After the intervention is completed, the qualitative component of the study will be carried out to access of the users' acceptability and satisfaction. It considers 12 semi-structured interviews to members of the EG group. The maximum variation sampling strategy will be used according to the completion of the intervention. An open coding of Grounded Theory will be used to data analysis.

The feasibility of m-health version of WWWT will be evaluated in terms of eligibility rates, recruitment rates and reasons for study refusals, feasibility to deliver the three components of the intervention, data attrition and follow-up rates by treatment condition. Their acceptability considers participant completion of the intervention rates, and a qualitative assessment of the users' acceptability and satisfaction. Quantitative indicators of feasibility and acceptability will be presented on frequency and/or percentage. Secondary outcomes will include: changes in maternal postnatal symptoms of depression and anxiety, change in parenting self-efficacy and perceived social support in both groups. Mixed-ANOVA analysis will be used to examine this variables differences between EG and CG whilst subjecting participants to repeated measures.

ELIGIBILITY:
Inclusion Criteria:

* First time mothers
* Adult (18 -64 years old)
* Having a healthy infant who is 6-8 weeks age
* Receive medical care in a primary health centers
* Having access to a mobile phone with instant messaging services (i.e., Whatsapp)
* Fluent in Spanish

Exclusion Criteria:

* Severe mental health problem (i.e. schizophrenia, mood disorder with suicidal ideation)
* Cognitive disability
* Actual substance abuse
* High risk for presenting symptoms of depression (EPDS above cut-off score)
* Severe psychosocial problem (i.e. domestic violence, sexual abuse).

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women is selected, since only they have the biological capacity to have children
Enrollment: 90 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Eligibility rate as feasibility indicator | At the baseline assessment during the recruitment period.
  Proportion of women who meet inclusion criteria compared with the total number of new mothers registered during the recruitment period in each participating primary health center
Recruitment rate as feasibility indicator | At the baseline assessment during the recruitment period.
  Proportion of mothers who accept the invitation to participate in the study respect to those meet eligibility criteria
Percentage of EG participants who receive the 12 psychoeducational modules, who attend the virtual meeting and who -at least- once established contact with the program facilitator | At 4-weeks from beginning intervention (when intervention finished)
  The feasibility to deliver the components of the intervention will be measured in terms of the percentage of participants of the EG who receive the 12 psychoeducational modules, who attend the virtual meeting and who -at least- once established contact with the program facilitator.
Percentage of participants who finished intervention by group as acceptability indicator | At 4-weeks from beginning intervention (when intervention finished).
  Proportion of participants who finished the intervention compared with a number of participant who began intervention in each group
Percentage of participant retention at follow-up by group as acceptability indicator | At 12-weeks after the completion of the intervention (follow-up measurement).
  Proportion of participants who remain in the study at the 12 weeks follow up compared with a number of participant who began intervention in each group

SECONDARY OUTCOMES:
Changes in maternal postnatal symptoms of depression, according to mean scores obtained with the Edinburgh Postnatal Depression Scale (EPDS) | At baseline (a week before the intervention starts) and 12-weeks after the completion of the intervention (follow-up measurement).
  The EPDS is a 10-item, self-report questionnaire used for screening current maternal symptoms of depression using a 4-point scale, total score ranging from 0 to 30 points. This scale has been validated in Chile.
Change in maternal postnatal symptoms of anxiety according to mean scores obtained with the Perinatal Anxiety Screening Scale (PASS) | At baseline (a week before the intervention starts) and 12-weeks after the completion of the intervention (follow-up measurement).
  The PASS is a 31-item, self-report questionnaire assesses maternal perinatal anxiety over the past month. A total score is calculated by adding all items that indicates level of severity: minimal (0-20 points), mild to moderate (21-41 points) and severe (42-93). The PASS includes four subscales, namely general worry and specific fears; perfectionism, control and trauma; social anxiety; and acute anxiety and adjustment.
Changes on perceived social support according to mean scores obtained with the multidimensional perceived social support scale (MSPSS) | At baseline (a week before the intervention starts) and 12-weeks after the completion of the intervention (follow-up measurement).
  The MSPSS is a 12 items self-report scale. It includes 3 subscales on perceived social support in three areas: family, friends and significant. Each item is rated on a 7-point Likert-scale (1 = very strongly disagree; 7 = very strongly agree). Three subscales' scores (range 4 to 28) and a total score (range 12 to 84) are estimated by adding the item scores. It has been translated and validated for the Chilean population.
Change in maternal self-efficacy according to mean scores obtained with the Parental Evaluation Scale (PEE) | At baseline (a week before the intervention starts) and 12-weeks after the completion of the intervention (follow-up measurement).
  The PEE is a 10-items self-report questionnaire to assess satisfaction and self-efficacy feelings about motherhood in women with children ages 0-2 years. Each item is rated on a 11-point scale (0=strongly disagree; 10=strongly agree) and the total score is estimated by adding item scores and then divided by 10

OTHER OUTCOMES:
Reasons for study refusals as a feasibility indicator | At the baseline assessment during the recruitment period.
  A list will be made containing the different reasons given by women who refused to participate, the results will be aggregated in terms of percentages.
Acceptability and satisfaction of the intervention from EG mothers' perspective | During a 12 weeks period following the completion of the intervention
  EG mothers' acceptability and satisfaction with the intervention, assessed through qualitative semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Soledad Coo, Principal Investigator — Universidad del Desarrollo
Locations (2):
- Chile (2):
  - Primary Health Center San Luis, Santiago, RMN
  - Primary Health Center Cardenal Silva Henríquez, Santiago, RM

IPD SHARING:
Plan to Share IPD: Yes
Individual quantitative participant data that underlie the reported results, after deidentification (text, tables and figures).
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: These data will be available to researchers who provide a methodologically sound proposal for the purposes of achieving specific aims outlined in that proposal. Proposals should be directed to Soledad Cood and J. Carola Pérez via email (scoo@udd.cl; janetperez@udd.cl) and will be reviewed by both researchers. Requests to access data to undertake hypothesis-driven research will not be unreasonably withheld. To gain access, data requesters will need to sign a data access agreement and to confirm that data will only be used for the agreed purpose for which access was granted and this these data will be not shared to other people.

REFERENCES:
- [Derived] Perez JC, Aldoney D, Garcia MI, Olhaberry M, Fernandez O, Alamo N, Franco P, Perez F, Fisher J, Rowe H, Coo S. Online intervention to prevent postnatal depression and anxiety in Chilean new mothers: Protocol for a feasibility trial. Health Informatics J. 2022 Oct-Dec;28(4):14604582221135440. doi: 10.1177/14604582221135440. PMID 36300324